CLINICAL TRIAL: NCT00830336
Title: A Relative Bioavailability Study of 200mg/5 mL Azithromycin Oral Suspension Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R05-1375
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Azithromycin; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azithromycin (test) (Experimental): Azithromycin for Oral Suspension 200 mg/5 mL (test) dosed in first period followed by Zithromax® Oral Suspension 200 mg/5 mL (reference) dosed in second period
  Interventions: Drug: Azithromycin
- Zithromax® (reference) (Active Comparator): Zithromax® for Oral Suspension 200 mg/5 mL (reference) dosed in first period followed by Azithromycin for Oral Suspension 200 mg/5 mL (test) dosed in second period
  Interventions: Drug: Zithromax®

INTERVENTIONS:
Drug: Azithromycin — Oral Suspension
  Arms: Azithromycin (test)
Drug: Zithromax® — Oral Suspension
  Other Names: Zithromax® for Oral Suspension
  Arms: Zithromax® (reference)

SUMMARY:
The study will compare the relative bioavailability (rate and extent of absorption) of 200 mg/5 mL Azithromycin oral suspension manufactured by TEVA Pharmaceutical Industries Ltd.; distributed by TEVA Pharmaceuticals USA with that of 200 mg/5 mL ZITHROMAX oral suspension distributed by Pfizer labs, a division of Pfizer Inc. following a single oral 10 mL dose (400 mg) in healthy adult subjects administered under non-fasting conditions.

DETAILED DESCRIPTION:
Detailed Description

Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

Outcome: Confidence interval fell within 80-125% therefore met the FDA Bioequivalence criteria; no drug related, serious, unexpected adverse events were reported during the study.

ELIGIBILITY:
Inclusion Criteria

* Screening Demographics: All subjects selected for this study will be healthy men and women 18 years of age or older at the time of dosing. The subject's body mass index (BMI) should be between 19 and 30.
* Screening Procedures: Each subject will complete the screening process within 28 days prior to period I dosing.
* Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed and signed by each potential participant before full implementation of screening procedures.
* Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature.
* The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.
* The screening clinical laboratory procedures will include:

  * HEMATOLOGY: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count
  * CLINICAL CHEMISTRY: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase
  * HIV antibody, hepatitis GB surface antigen, hepatitis C antibody screens
  * URINALYSIS: by dipstick; full microscopic examination if dipstick positive
  * URINE DRUG SCREEN: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine
  * SERUM PREGNANCY SCREEN (female subjects only)
* If female and:

  * Of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condom with spermicide, diaphragm with spermicide, intrauterine device (IUD), or abstinence; or
  * Is postmenopausal for at least 1 year; or
  * Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) Exclusion Criteria
* Subjects with a recent history of drug or alcohol addiction or abuse.
* Subjects with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Subjects whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Subjects demonstrating a reactive screen for hepatitis B surface antigen, hepatitis C antibody or HIV antibody.
* Subjects demonstrating a positive drug abuse screen when screened for this study.
* Female subjects demonstrating a positive pregnancy screen.
* Female subjects who are currently breastfeeding.
* Subjects with a history of allergic response(s) to azithromycin or related drugs.
* Subjects with a history of clinically significant allergies including drug allergies.
* Subjects with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Subjects who currently or report using tobacco products within 90 days of Period I dose administration.
* Subjects who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
* Subjects who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Subjects who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Subjects who report receiving any investigational drug within 28 days prior to Period I dosing.
* Subjects who report taking any systemic prescription medication in the 14 days prior to Period I dosing.
* Subjects who report an intolerance of direct venipuncture.
* Subjects who report consuming an abnormal diet during the 28 days prior to Period I dosing.
* Female subjects who report using implanted or injected hormonal contraceptives (birth control) during the 6 months prior to Period I dosing.
* Female subjects who report using oral hormonal contraceptives (birth control) during the 14 days prior to Period I dosing.
* Subjects who report having difficulty fasting or consuming standardized meals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute Ltd., Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin (Test) First: Azithromycin for Oral Suspension 200 mg/5 mL (test) dosed in first period followed by Zithromax® Oral Suspension 200 mg/5 mL (reference) dosed in second period
- Zithromax® (Reference) First: Zithromax® for Oral Suspension 200 mg/5 mL (reference) dosed in first period followed by Azithromycin for Oral Suspension 200 mg/5 mL (test) dosed in second period
Period: First Intervention
Arm/Group | Azithromycin (Test) First | Zithromax® (Reference) First
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0
Period: Washout: 21 Days
Arm/Group | Azithromycin (Test) First | Zithromax® (Reference) First
Started | 40 | 40
Completed | 39 | 40
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Azithromycin (Test) First | Zithromax® (Reference) First
Started | 39 | 40
Completed | 39 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin (Test) First | Zithromax® (Reference) First | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 39 | 78
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 44
  Male | 21 | 15 | 36
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 37 | 37 | 74
  Black | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native American | 0 | 2 | 2
  Pacific Islander/Hawaiian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 168 hour period
Population: Samples for two subjects who completed the study were not analyzed per protocol due to emesis during the sample collection period.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Azithromycin: Azithromycin for Oral Suspension 200 mg/5 mL (test) dosed in either period
- Zithromax®: Zithromax® for Oral Suspension 200 mg/5 mL (reference) dosed in either period
Arm/Group | Azithromycin | Zithromax®
Number analyzed (Participants) | 77 | 77
ng/mL | 560.56 (212.71) | 562.97 (254.40)
Statistical Analysis 1: Comparison: Azithromycin vs Zithromax®; Test type: Non-Inferiority or Equivalence — The pharmacokinetic parameters were evaluated statistically by an analysis of variance (ANOVA) appropriate for the experimental design of this study; Geometric Test/Ref Ratio x 100 = 103.08, 90% CI [95.41 to 111.37] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 168 hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Azithromycin | Zithromax®
Number analyzed (Participants) | 77 | 77
ng*h/mL | 5140.47 (1630.93) | 4884.55 (1599.27)
Statistical Analysis 1: Comparison: Azithromycin vs Zithromax®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Test/Ref Ratio x 100 = 105.84, 90% CI [99.33 to 112.77] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 168 hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Azithromycin | Zithromax®
Number analyzed (Participants) | 77 | 77
ng*h/mL | 4555.91 (1502.93) | 4277.83 (1431.90)
Statistical Analysis 1: Comparison: Azithromycin vs Zithromax®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Test/Ref Ratio x 100 = 107.04, 90% CI [99.96 to 114.62] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.